CLINICAL TRIAL: NCT00143975
Title: Phase II Study on Gemtuzumab Ozogamicin in Combination With All-trans-Retinoic Acid, High-dose Cytarabine and Mitoxantrone in Patients With Primary Refractory Acute Myeloid Leukemia
Brief Title: Gemtuzumab Ozogamicin in Combination With A-HAM in Refractory AML (GO-A-HAM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Prof. Dr. Reinhard Marre, University of Ulm
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG05-04
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute myeloid leukemia; gemtuzumab ozogamicin; refractory disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Disease | interventions — Cytarabine; Mitoxantrone; Gemtuzumab

INTERVENTIONS:
Drug: Cytarabine — 3 g/m2 bid. i.v day 1-3
Drug: Mitoxantrone — 12 mg/m2 i.v. day 2 and 3
Drug: Gemtuzumab Ozogamicin — 3mg/m² i.v. day 1
Drug: All-trans-Retinoid Acid — 45 mg/m2 p.o. day 4-6 15 mg/m2 p.o. day 7-28

SUMMARY:
GO-A-HAM:

Gemtuzumab Ozogamicin 3g/m² day 1 Cytarabine 3g/m² bid days 1-3 Mitoxantrone 12mg/m² days 2,3 All-trans Retinoic acid 45mg/m² days 4-6 and 15 mg/m² days 7-28

DETAILED DESCRIPTION:
Primary refractory AML is associated with an extremely poor prognosis [1,2]. In the AMLHD93 trial conducted by the AMLSG ULM, patients refractory to the first induction therapy with ICE (idarubicin, cytarabine, etoposide) had an overall survival of 12% after 5 years [1]. All patients alive in this cohort had received allogeneic transplantation. Therefore, we assigned allogeneic transplantation in our consecutive trial, AMLHD98A, to all primary refractory patients [3]. However, the main problem in this patient group remains achieving a partial (PR) or complete (CR) remission to a salvage therapy. Additionally, the pre-transplant disease status is an important prognostic factor in most studies of allogeneic transplantation, regardless dose intensified or dose reduced conditioning regimens are used [4,5,6]. Since 1993, in all studies of the German-Austrian-AMLSG response-adapted treatment strategies had been used. Within the AMLHD93 trial, refractory patients were assigned to an intensified second induction regimen with S-HAM (age<55 years) [7] or HAM (age 55 to 60 years) [1], and in the AMLHD98A trial, with A-HAM [3]. The incorporation of all-trans-retinoic acid was based on in vitro data [8-13] and by our randomised AMLHD98B study for elderly AML-patients showing a benefit in primary response and survival for patients assigned to standard induction therapy in combination with ATRA [14].

To compare the different salvage therapy strategies, we performed an as-treated analysis in primary refractory patients of the different cohorts. Although refractory to the first induction therapy with ICE, nine patients received a second cycle ICE. The results summarized in table 1 showed an improved response rate (CR and PR) for patients treated with the A-HAM protocol and thus leading to a higher proportion of patients receiving an allogeneic transplantation. Survival analysis showed so far no difference between the 4 different groups. Gemtuzumab ozogamicin (GO) is a humanized anti-CD33 conjugated to Calicheamicin. The efficacy and the toxicity profile has been evaluated in several studies, so far the substance is approved for the monotherapy in relapsed AML-patients in a dose of 9mg/m² q 14d [15]. However, used as a single agent the efficacy is limited and not durable. Therefore, several trials have evaluated GO in combination with conventional chemotherapy [16,17]. In the MRC study a dose of 6 mg/m² given once at day 1 was associated with an increased liver toxicity and therefore the study continues with a dose of 3 mg/m² once at day 1 of induction therapy [17]. In summary, the available data for combination therapy showed efficacy of GO in phase II trials. The dose limiting toxicity was defined in the MRC trial at 6 mg/m². Therefore we consider GO in combination with A-HAM for primary refractory adult AML patients. Because all primary refractory patients are candidates for an allogeneic transplantation special considerations have to be taken with respect to the development of VOD after allogeneic transplantation. One recent report suggests a substantial risk for VOD for patients receiving an allogeneic transplantation after a therapy with GO [18]. In this report the odds ratio for VOD after a therapy with GO within 3.5 months before allogeneic transplantation was 21.6 (95%-confidence interval 4.2-112.2%). However, this report is based on 62 patients and the dosage of GO used was 6mg/m² and 9mg/m². Therefore, holding in mind the risk of VOD after GO exposure and the extremely poor prognosis of primary refractory patients the treatment approach combining A-HAM with GO with a dose of 3mg/m² is justified.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia defined according the WHO classification not responding to first induction therapy
* Age 18-60 years
* Written informed consent

Exclusion Criteria:

* Acute promyelocytic leukemia
* Uncontrolled infection
* Transfusion-refractory thrombocytopenia
* Pregnancy, breast-feeding, insufficient contraception
* Organ insufficiency: kidneys, liver, lungs, heart
* Severe neurological and psychiatrical interfering with informed consent
* No consent for the registration, storage and processing of data concerning the characteristics of the AML and the individual course
* Performance status > grad 2 according the WHO classification

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2004-06; Primary Completion 2007-07 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
CR-rate after therapy with GO-A-HAM | day 30

SECONDARY OUTCOMES:
kind, incidence, severity, temporal sequence and correlation of side effects of the study-drugs | 30 days
rate of veno occlusive disease (VOD) after allogene transplantation | 100 days after allogene transplantation
overall survival | two years

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Schlenk, Dr. med., Principal Investigator — University of Ulm / Department of Internal Medicine III
Locations (27):
- Austria (3):
  - Department of Hematology / Oncology, University Hospital of Innsbruck, Innsbruck
  - St. Johann Hospital, Clinical Center of Salzburg, Salzburg
  - Medical Department III, Hanusch-Hospital, Vienna
- Germany (24):
  - Medical Department II, Central Hospital of Augsburg, Augsburg
  - Department of General Internal Medicine, University Hospital of Bonn, Bonn
  - Department of Hematology and Oncology, Hospital Essen-Süd, Ev. Hospital of Essen-Werden, Essen
  - Department of Internal Medicine III, City Hospital Frankfurt am Main - Höchst, Frankfurt
  - Medical Department IV, University Hospital of Gießen, Giessen
  - Department of Internal Medicine, Wilhelm-Anton-Hospital gGmbH, Goch
  - Centre of Internal Medicine, University Hospital of Göttingen, Göttingen
  - Department of Oncology and Hematology, University Hospital Eppendorf, Hamburg
  - Medical Department III, Clinical Center Hanau, Hanau
  - Medical Department III, Clinical Center Hannover-Siloah, Hanover
  - Department of Hematology, Hemostaseology and Oncology, Medizinische Hochschule Hannover, Hanover
  - Department of Internal Medicine I, University Hospital of Saarland, Homburg
  - Medical Department II, City Hospital Karlsruhe gGmbH, Karlsruhe
  - Medical Department II, University Hospital of Kiel, Kiel
  - Department of Internal Medicine / Hematology and Oncology, Caritas Hospital Lebach, Lebach
  - Department of Hematology / Oncology, Clinical center of Lüdenscheid, Lüdenscheid
  - Department of Hematology and internal Oncology, University Hospital of Mainz, Mainz
  - Medical Department III, Clinical Center rechts der Isar, München
  - Department of Hematology and Oncology, Clinical Center of Oldenburg gGmbH, Oldenburg
  - Department of Hematology and Oncology / Caritas Hospital St. Theresia, Saarbrücken
  - Department of Oncology / Clinical Center of Stuttgart, Stuttgart
  - Department of Internal Medicine II, University Hospital of Tübingen, Tübingen
  - Department of Internal Medicine III, University of Ulm, Ulm
  - Medical Department I, Helios Hospital Wuppertal, Wuppertal

REFERENCES:
- [Background] Schlenk RF, Benner A, Hartmann F, del Valle F, Weber C, Pralle H, Fischer JT, Gunzer U, Pezzutto A, Weber W, Grimminger W, Preiss J, Hensel M, Frohling S, Dohner K, Haas R, Dohner H; AML Study Group Ulm (AMLSG ULM). Risk-adapted postremission therapy in acute myeloid leukemia: results of the German multicenter AML HD93 treatment trial. Leukemia. 2003 Aug;17(8):1521-8. doi: 10.1038/sj.leu.2403009. PMID 12886238
- [Background] Wheatley K, Burnett AK, Goldstone AH, Gray RG, Hann IM, Harrison CJ, Rees JK, Stevens RF, Walker H. A simple, robust, validated and highly predictive index for the determination of risk-directed therapy in acute myeloid leukaemia derived from the MRC AML 10 trial. United Kingdom Medical Research Council's Adult and Childhood Leukaemia Working Parties. Br J Haematol. 1999 Oct;107(1):69-79. doi: 10.1046/j.1365-2141.1999.01684.x. PMID 10520026
- [Background] Schlenk RF, Fröhling S, Del Valle F, Dreger P, Fischer JTh, Glasmacher A, Götze K, Grimminger W, Germing U, Hartmann F, Koller E, Mergenthaler HG, Salwender H, Waterhouse C, Döhner K, Bunjes D, Döhner H. Early Allogeneic Transplantation in Patients with High Risk Acute Myeloid Leukemia Defined by Karyotype and Response To Induction Therapy: First Results of the AML HD98A Trial. Blood 98: 2822, abstract
- [Background] Bunjes D, Buchmann I, Duncker C, Seitz U, Kotzerke J, Wiesneth M, Dohr D, Stefanic M, Buck A, Harsdorf SV, Glatting G, Grimminger W, Karakas T, Munzert G, Dohner H, Bergmann L, Reske SN. Rhenium 188-labeled anti-CD66 (a, b, c, e) monoclonal antibody to intensify the conditioning regimen prior to stem cell transplantation for patients with high-risk acute myeloid leukemia or myelodysplastic syndrome: results of a phase I-II study. Blood. 2001 Aug 1;98(3):565-72. doi: 10.1182/blood.v98.3.565. PMID 11468151
- [Background] Schlenk RF, Hartmann F, Hensel M, Jung W, Weber-Nordt R, Gabler A, Haas R, Ho AD, Trumper L, Dohner H. Less intense conditioning with fludarabine, cyclophosphamide, idarubicin and etoposide (FCIE) followed by allogeneic unselected peripheral blood stem cell transplantation in elderly patients with leukemia. Leukemia. 2002 Apr;16(4):581-6. doi: 10.1038/sj.leu.2402423. PMID 11960336
- [Background] Sierra J, Storer B, Hansen JA, Martin PJ, Petersdorf EW, Woolfrey A, Matthews D, Sanders JE, Storb R, Appelbaum FR, Anasetti C. Unrelated donor marrow transplantation for acute myeloid leukemia: an update of the Seattle experience. Bone Marrow Transplant. 2000 Aug;26(4):397-404. doi: 10.1038/sj.bmt.1702519. PMID 10982286
- [Background] Hiddemann W, Buchner T, Essink M, Koch O, Stenzinger W, van de Loo J. High-dose cytosine arabinoside and mitoxantrone: preliminary results of a pilot study with sequential application (S-HAM) indicating a high antileukemic activity in refractory acute leukemias. Onkologie. 1988 Feb;11(1):10-2. doi: 10.1159/000216471. PMID 3283619
- [Background] Hu ZB, Minden MD, McCulloch EA. Direct evidence for the participation of bcl-2 in the regulation by retinoic acid of the Ara-C sensitivity of leukemic stem cells. Leukemia. 1995 Oct;9(10):1667-73. PMID 7564507
- [Background] Bradbury DA, Aldington S, Zhu YM, Russell NH. Down-regulation of bcl-2 in AML blasts by all-trans retinoic acid and its relationship to CD34 antigen expression. Br J Haematol. 1996 Sep;94(4):671-5. doi: 10.1046/j.1365-2141.1996.d01-1838.x. PMID 8826891
- [Background] Benito A, Grillot D, Nunez G, Fernandez-Luna JL. Regulation and function of Bcl-2 during differentiation-induced cell death in HL-60 promyelocytic cells. Am J Pathol. 1995 Feb;146(2):481-90. PMID 7856757
- [Background] Yang GS, Minden MD, McCulloch EA. Influence of schedule on regulated sensitivity of AML blasts to cytosine arabinoside. Leukemia. 1993 Jul;7(7):1012-9. PMID 7686602
- [Background] Zheng A, Mantymaa P, Saily M, Savolainen E, Vahakangas K, Koistinen P. p53 pathway in apoptosis induced by all-trans-retinoic acid in acute myeloblastic leukaemia cells. Acta Haematol. 2000;103(3):135-43. doi: 10.1159/000041036. PMID 10940651
- [Background] Schlenk RF, Frohling S, Hartmann F, Fischer JT, Glasmacher A, del Valle F, Grimminger W, Gotze K, Waterhouse C, Schoch R, Pralle H, Mergenthaler HG, Hensel M, Koller E, Kirchen H, Preiss J, Salwender H, Biedermann HG, Kremers S, Griesinger F, Benner A, Addamo B, Dohner K, Haas R, Dohner H; AML Study Group Ulm. Phase III study of all-trans retinoic acid in previously untreated patients 61 years or older with acute myeloid leukemia. Leukemia. 2004 Nov;18(11):1798-803. doi: 10.1038/sj.leu.2403528. PMID 15385923
- [Background] Sievers EL, Larson RA, Stadtmauer EA, Estey E, Lowenberg B, Dombret H, Karanes C, Theobald M, Bennett JM, Sherman ML, Berger MS, Eten CB, Loken MR, van Dongen JJ, Bernstein ID, Appelbaum FR; Mylotarg Study Group. Efficacy and safety of gemtuzumab ozogamicin in patients with CD33-positive acute myeloid leukemia in first relapse. J Clin Oncol. 2001 Jul 1;19(13):3244-54. doi: 10.1200/JCO.2001.19.13.3244. PMID 11432892
- [Background] De Angelo, D., et al., Interim analysis of a phase II study of the safety and efficacy of Gemtuzumab Ozogamicin (Mylotarg) given in combination with Cytarabine and Daunorubicin in patients< 60years old with untreated acute myeloid leukemia. Blood 100:745a.
- [Background] Jonathan W. Kell, Alan K. Burnett, Raj Chopra, John Yin, Dominic Culligan, Richard Clark, Ann Hunter, Ama Rohatiner, Don W. Milligan, Nigel Russell, Archie Prentice. Dept of Haematology, MRC AML Pilot Group, United Kingdom Mylotarg (Gemtuzumab Ozogamicin: GO) Given Simultaneously with Intensive Induction and/or Consolidation Therapy for AML Is Feasible and May Improve the Response Rate. Blood 100:746a
- [Background] Wadleigh M, Richardson PG, Zahrieh D, Lee SJ, Cutler C, Ho V, Alyea EP, Antin JH, Stone RM, Soiffer RJ, DeAngelo DJ. Prior gemtuzumab ozogamicin exposure significantly increases the risk of veno-occlusive disease in patients who undergo myeloablative allogeneic stem cell transplantation. Blood. 2003 Sep 1;102(5):1578-82. doi: 10.1182/blood-2003-01-0255. Epub 2003 May 8. PMID 12738663
- [Derived] Hutter-Kronke ML, Benner A, Dohner K, Krauter J, Weber D, Moessner M, Kohne CH, Horst HA, Schmidt-Wolf IG, Rummel M, Gotze K, Koller E, Petzer AL, Salwender H, Fiedler W, Kirchen H, Haase D, Kremers S, Theobald M, Matzdorff AC, Ganser A, Dohner H, Schlenk RF. Salvage therapy with high-dose cytarabine and mitoxantrone in combination with all-trans retinoic acid and gemtuzumab ozogamicin in acute myeloid leukemia refractory to first induction therapy. Haematologica. 2016 Jul;101(7):839-45. doi: 10.3324/haematol.2015.141622. Epub 2016 Apr 1. PMID 27036160